CLINICAL TRIAL: NCT04897698
Title: LB001 Study: Probiotics for Weight Loss: A Randomized Controlled Study
Brief Title: Probiotics for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: deFair Medical AB (Unknown)
Responsible Party: Principal Investigator, Emilia Hagman, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-1326/2021
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Four capsules containing rice flour will be given to the placebo group daily.
  Interventions: Dietary Supplement: LB001
- Single dose (Experimental): Two capsules of probiotics and two capsules of placebo daily. Probiotic capsules contains strains of pediococcus (Bacterial family of Lactobacillaceae) and saccharomycetes (kingdom of Fungi and the division Ascomycota) with a concentration of 13 millions cfu/g. Other ingredients (including stabilization) include rice bran, vegetable L-Cystein, magnesium salts from vegetable fatty acids. The capsule shell is made of vegetable HydroxyPropylMetylCellulosa (HPMC). Each capsule has a weight of 0.4 gram.
  The placebo is made of rice flour.
  Interventions: Dietary Supplement: LB001
- Double dose (Experimental): Four capsules of probiotics daily. Probiotic capsules contains strains of pediococcus (Bacterial family of Lactobacillaceae) and saccharomycetes (kingdom of Fungi and the division Ascomycota) with a concentration of 13 millions cfu/g. Other ingredients (including stabilization) include rice bran, vegetable L-Cystein, magnesium salts from vegetable fatty acids. The capsule shell is made of vegetable HydroxyPropylMetylCellulosa (HPMC). Each capsule has a weight of 0.4 gram.
  Interventions: Dietary Supplement: LB001

INTERVENTIONS:
Dietary Supplement: LB001 — Probiotics

SUMMARY:
This study will investigate a compound of probiotics and prebiotics in females and males with overweight with the aim to evaluate the effect on weight and metabolic markers.

The design is a three month randomized doubled-blinded, three-armed placebo-controlled trial of probiotics for weight loss. Normal dose (2 capsules á 0.4g per day) doubled dose (4 capsules á 0.4g per day), or placebo.

A second, non-blinded, phase with only the compound of probiotics and prebiotics, with tripple dose (6 capsuled á 0.4g per day), will be performed for individuals who had the compound in the first phase.

DETAILED DESCRIPTION:
Participants Total number of study participants will be 75-90, consisting of overweight men and women, 18-45 years of age.

Treatment Dietary supplement consisting of probiotic capsules called LB001. It contains strains of pediococcus (Bacterial family of Lactobacillaceae) and saccharomycetes (kingdom of Fungi and the division Ascomycota) with a concentration of 13 millions cfu/g. Other ingredients (including stabilization) include rice bran, vegetable L-Cystein, magnesium salts from vegetable fatty acids. The capsule shell is made of vegetable HydroxyPropylMetylCellulosa (HPMC). Each capsule has a weight of 0.4 gram. The placebo is made of rice flour.

Since one of the inclusion criteria is "willingness to lose weight", all study participants, regardless of randomized treatment, will receive general advice regarding healthy lifestyle habits.

ELIGIBILITY:
Inclusion Criteria:

* BMI 26.0 - 29,99 kg/m2
* 18-45 years old
* Willingness to lose weight

Exclusion Criteria:

* Active weight loss in the last three months
* The desire for or planned pregnancy upcoming months
* Chronic somatic diseases that may affect metabolic and/or intestinal function (e.g. diabetes, hypertension, dyslipidemia, Irritable Bowel Disorder (IBD), gluten intolerance, pancreatic dysfunction, other causes of malabsorption, neoplastic disease)
* Allergies with previous anaphylactic reactions
* Abdominal surgery six months prior to inclusion
* Current or history of eating disorders
* Extreme or unusual diets for the last three months, which the investigator considers could negatively affect the outcome of the study
* Psychiatric disorders (e.g., schizophrenia, and other diagnoses that may influence compliance)
* Drug or alcohol abuse
* Continuous oral pharmacological treatment and other types of pharmacological treatment that may influence the study
* Present or recent usage of other probiotic agents
* Other conditions which the investigator considers could negatively affect the outcome of the study or study compliance

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2021-10-16 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Weight change | Baseline, 3-month follow-up
  Weight will be measured in kilograms using a scale.
Weight change | Baseline, 6-month follow-up
  Weight will be measured in kilograms using a scale.

SECONDARY OUTCOMES:
Waist circumference | Baseline, 3-month follow-up
  Participants waist circumference will be measured using a standard tape measure (in cm).
Waist circumference | Baseline, 6-month follow-up
  Participants waist circumference will be measured using a standard tape measure (in cm).
HbA1c | Baseline, 3-month follow-up
  Glycated hemoglobin A1c will be measured in blood (mmol/mol)
HbA1c | Baseline, 6-month follow-up
  Glycated hemoglobin A1c will be measured in blood (mmol/mol)
HDL | Baseline, 3-month follow-up
  High-density lipoproteins will be measured in plasma (mmol/L)
HDL | Baseline, 6-month follow-up
  High-density lipoproteins will be measured in plasma (mmol/L)
Triglycerides | Baseline, 3-month follow-up
  Triglycerides will be measured in plasma (mmol/L)
Triglycerides | Baseline, 9-month follow-up
  Triglycerides will be measured in plasma (mmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Hagman, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Department of Clinical Science, Intervention and Technology, Huddinge, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Danielsson P, Putri RR, Marcus C, Hagman E. Evaluating probiotic efficacy on weight loss in adults with overweight through a double-blind, placebo-controlled randomized trial. Sci Rep. 2023 Oct 24;13(1):18200. doi: 10.1038/s41598-023-45395-7. PMID 37875559